CLINICAL TRIAL: NCT05592041
Title: In-vitro and Randomized Controlled Clinical Studying of Natural Constituents' Anti-HPV Potential for Treatment of Plantar Warts Supported With in Silico Studies
Brief Title: Studying of Natural Constituents' Treatment of Plantar Warts
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Principal Investigator, Soad Ali, lecturer of pharmaceutics and clinical pharmacy Deraya university, Deraya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anti-HPV
Record Dates: First submitted 2022-10-17; First posted 2022-10-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Plantar Wart

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Group I) (Experimental)
  Interventions: Drug: Banaba Leaf Extract
- Control group (Group II) (No Intervention)

INTERVENTIONS:
Drug: Banaba Leaf Extract — a herbal extract in the form of Bigel
  Other Names: moringa banna nigella
  Arms: Treatment group (Group I)

SUMMARY:
Moringa banana nigella and Banna coat extract were prepared and formulated in the form of bi gel for transdermal delivery of these plant extracts. The formulation was prepared and charterized for organoleptic charters, morphology, and penetration efficacy. The optimised formulation was assessed clinically on patients suffering from plantar warts. The clinical study was phase 1 and interventional randomised allocation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged 18 years or more.
* Clinical evaluation
* Number of warts lower than 10 on the 2 feet and total diameter of warts lower than 10 cm

Exclusion Criteria:

* Patient suspected to be immunocompromised
* Patient aged under 18 years
* Patient refusing to sign the consent
* Pregnant or lactating women

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Complete clinical remission of the warts | 30 days
  Number of warts (counts)
Clinical assessment of warts curement | 30 days
  Diameter of wart in cm

SECONDARY OUTCOMES:
Pain asssesment | 30 days
  pain was assesed by VAS scoring (0) the least to (5) highest

CONTACTS AND LOCATIONS:
Locations (1):
- Soad A. Mohamad, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided